CLINICAL TRIAL: NCT05284175
Title: A Prospective, Self-controlled Study to Explore Efficacy and Safety of Orelabrutinib in AQP4-IgG Positive Neuromyelitis Optica Spectrum Disorder
Brief Title: A Study of Orelabrutinib in Patients With AQP4-IgG Positive Neuromyelitis Optica Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing InnoCare Pharma Tech Co., Ltd. (Industry); GCP ClinPlus Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Yan Xu, Chief Physician, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-022-006
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica Spectrum Disorder; BTK inhibitors; Orelabrutinib
MeSH Terms: conditions — Neuromyelitis Optica | interventions — orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Orelabrutinib, orally, 50 mg QD (Experimental): Orelabrutinib, orally, 50 mg QD
  Interventions: Drug: Orelabrutinib

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib, orally, 50 mg QD

SUMMARY:
Neuromyelitis optica spectrum disorder (NMOSD) is a chronic inflammatory demyelinating autoimmune disease of the central nervous system. NMOSD is a highly relapsing, severely disabling disease. AQP4-IgG positive NMOSD is related to a specific aquaporin 4 antibody (AQP4 IgG) produced by mature B cells. BTK is a key kinase in B cell receptor signal transduction pathway. Abnormal activation of BTK related signaling pathway can lead to autoantibody production and autoimmune diseases. Therefore, BTK can be developed as a new target for autoimmune diseases.

DETAILED DESCRIPTION:
Approximately 23 subjects will be enrolled.

Experimental drug treatment: Orelabrutinib, 50mg, orally, once a day.

The subject will come to visit at week 0, 1, 2, 4, 8, 12, 16, 20, 24, 36, 48 and safety follow up visit which is planed 28 days after last administration.

Baseline patient assessment:

1. Baseline examination: vital signs, physical examination, blood routine examination, urine routine examination, liver and kidney function, coagulation function, thyroid function, HIV, HCV, HBV virus test, tuberculosis test, chest X-ray, ECG and pregnancy test.
2. Functional disability assessment: Expanded Disability Status Scale (EDSS) score and low contrast vision (LCVA) score.
3. EQ5D scale evaluation.
4. Serum AQP4-IgG titer, neuro filament light chain, T/B/NK cell count, Immunoglobulin (IgG, IgA and IgM)

ELIGIBILITY:
Inclusion Criteria:

* 1) 18-75 years old (inclusive) at the time of signing the informed consent form
* 2)Diagnosed with AQP4-IgG positive NMOSD in accordance with 2015 IPND diagnostic criteria.
* 3)Relapse ≥ 2 within 1 year before screening, and at least 1 relapse within 6 months before screening
* 4)If the subject has stable steroids treatment (≤ 7.5mg prednisone, or equivalent dose of steroids), the treatment needs to be stable more than 1 month before starting the study drug treatment.
* 5)EDSS ≤7.5 at screening
* 6)Negative pregnancy test for female of childbearing potential at screening
* 7)Understood the study procedure and voluntarily signed written informed consent

Exclusion Criteria:

* 1) History of serious heart, lung, liver, kidney, blood disease, etc.
* 2) Any major infection judged by the investigator requiring hospitalization and parenteral antimicrobial treatment within 1 month before screening
* 3) History of episodes of herpes zoster ≥ 2 or disseminated herpes zoster ≥ 1
* 4) History of or having any of the following medication / treatment: ① Received BTK inhibitor at any time in the past; ② B-cell targeted therapy within 12 weeks before the first dose; ③ Received biological agents within 12 weeks before the first dose; ④ Received live virus vaccine or live attenuated vaccine within 8 weeks before the first dose; ⑤ Received steroids treatment for other diseases within 6 months before screening, the dosage > 20mg / day for more than 21 days; ⑥ Used a study drug or other experimental treatment within 4 weeks before screening or 5 half-lives, or participating in any other intervention clinical trial.
* 5) During screening or baseline examination, laboratory results meet the exclusion criteria:

  * Human immunodeficiency virus (HIV) positive
  * Hepatitis C virus (HCV) antibody positive. (If a subject has a history of HCV infection, has completed and recorded appropriate treatment at least 1 year before screening, and the HCV RNA measured by PCR at the time of screening is negative, the subject will not be excluded from this study.)
  * Hepatitis B surface antigen (HBsAg) positive and / or hepatitis B core antibody (HBcAb) positive
  * Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2
  * ALT/AST > 2 x ULN, Total Bilirubin > 1.5 x ULN, or any other clinically significant laboratory abnormality
  * Neutrophil < 1500 / mm3, platelet < 75000 / mm3, lymphocyte < 1000 / mm3 or leukocyte < 3500 / mm3.
  * International standardized ratio (INR) ≥ 1.5 or activated partial thromboplastin time (APTT) ≥ 1.5x ULN.
  * CD19 B cells lower than the lower limit of the normal range
* 6) Used strong to medium CYP3A inducers within 3 weeks before treatment, or strong to medium CYP3A inhibitors within 1 week before treatment, or strong to medium CYP3A inducers or inhibitors may be used during treatment.
* 7) There are situations that other researchers think are not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Annualized relapse rate at week 48 compared with that before baseline. | week 48
  Annualized relapse rate at week 48 compared with that before baseline.

SECONDARY OUTCOMES:
Proportion of patients without relapse | weeks 24 and 48
  Proportion of patients without relapse at weeks 24 and 48;
Changes in the expanded disability status scale (EDSS) score from baseline | weeks 4, 12, 24, 36 and 48
  Changes in the expanded disability status scale (EDSS) score from baseline at weeks 4, 12, 24, 36 and 48;
Changes in low contrast visual acuity score (LCVA) from baseline | weeks 4, 12, 24, 36 and 48
  Changes in low contrast visual acuity score (LCVA) from baseline at weeks 4, 12, 24, 36 and 48;
Changes in EQ5D scores from baseline | weeks 12, 24, 36 and 48
  Changes in EQ5D scores from baseline at weeks 12, 24, 36 and 48;
Changes in serum AQP4-IgG titer and neurofilament light chain protein level from baseline | weeks 4, 12, 24, 36 and 48
  Changes in serum AQP4-IgG titer and neurofilament light chain protein level from baseline at weeks 4, 12, 24, 36 and 48;
Changes in absolute value of peripheral blood B cell count and immunoglobulin (IgA, IgM, IgG) from baseline | weeks 4, 12, 24, 36 and 48
  Changes in absolute value of peripheral blood B cell count and immunoglobulin (IgA, IgM, IgG) at weeks 4, 12, 24, 36 and 48 from baseline;
Percentage of patients who withdraw from the study due to adverse events. | weeks1, 2, 4, 8, 12, 16, 20, 24, 36 , 48
  Percentage of patients who withdraw from the study due to adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xu, Doctor, Principal Investigator — Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No